CLINICAL TRIAL: NCT02685930
Title: Pneumonia in the Intensive Care Unit (ICU) Setting
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Marin Kollef, M.D., FACP, FCCP, Professor of Medicine, Washington University School of Medicine
Other Study IDs: 201509075
Record Dates: First submitted 2016-01-26; First posted 2016-02-19 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Pneumonia; Respiratory Failure
Keywords: invasive mechanical ventilation
MeSH Terms: conditions — Pneumonia; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Microbiological: tracheal aspirate, bronchialalveolar lavage, blood cultures, viral PCR multiplex from respiratory specimen Bronchialalveolar lavage: Cell count and differential
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pneumonia without ICU stewardship involvement: Patients receiving >24 hours of invasive mechanical ventilation for pneumonia-related respiratory failure. Antibiotic choice and duration of therapy will not be influenced by the dedicated ICU stewardship team.
- Pneumonia with ICU stewardship involvement: Patients receiving >24 hours of invasive mechanical ventilation for pneumonia-related respiratory failure. Recommendations for antibiotic choice and duration of therapy will be provided by the dedicated ICU stewardship team (consisting of pulmonary fellows and ICU pharmacists)
  Interventions: Behavioral: Antibiotic de-escalation by ICU stewardship team with decreased exposure to broad spectrum antibiotics and shorter duration of therapy

INTERVENTIONS:
Behavioral: Antibiotic de-escalation by ICU stewardship team with decreased exposure to broad spectrum antibiotics and shorter duration of therapy — ICU stewardship team will provide recommendations to the ICU team regarding antibiotic de-escalation and duration of therapy in attempts of improving antibiotic stewardship practices without compromising patient outcomes.Recommendations will be based on patient showing clinical improvement combined with microbial culture data.
  Groups: Pneumonia with ICU stewardship involvement

SUMMARY:
The purpose of this observational study is to collect prospective data on the occurrence of bacterial and viral pneumonia in the ICU setting. Current classification systems for pneumonia promote over treatment with antibiotics as they do not specifically recognize the presence of culture-negative and viral pneumonia. The investigators will collect data to determine if a novel pneumonia classification system can be developed that more accurately links the etiology of pneumonia (antibiotic-susceptible bacterial pneumonia, antibiotic-resistant bacterial pneumonia, culture-negative pneumonia, viral pneumonia) to clinical outcomes. Additionally, the investigators will collect data on the practice of antimicrobial stewardship in the ICU setting to determine if further improvements in antibiotic practices can be accomplished in the future.

DETAILED DESCRIPTION:
The investigators will be prospectively collecting data on patients admitted to the 8300 and 8400 medical intensive care units at Barnes-Jewish Hospital requiring invasive mechanical ventilation for support in respiratory failure from pneumonia. Data will be collected on patients admitted from 1/2016-12/2016. The investigators will be collecting initial patient characteristic data as well as reviewing microbial specimen results (tracheal aspirate, bronchial alveolar lavage, viral multiplex, blood cultures) and antibiotic usage in real time. The investigators will identify any changes in antibiotic usage demonstrated with the advising of the ICU antibiotic stewardship team.

ELIGIBILITY:
Inclusion Criteria:

* age 18+, admitted for 8300 or 8400 medical ICU between 1/2016 and 12/2016 for respiratory failure from pneumonia, requirement of > 24 hours of invasive mechanical ventilatory support for pneumonia

Exclusion Criteria:

* Immunocompromised as defined by HIV/AIDS, known immunodeficiency, chronic steroids > 20mg/day Prednisone equivalent, other home immunosuppressants, solid organ or bone marrow transplant patients, cystic fibrosis, bronchiectasis, active malignancy, receiving chemotherapy or radiation therapy within the past 3 months, hematologic malignancy
* Chronic ventilator dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients in the 8300 and 8400 medical intensive care units at Barnes-Jewish Hospital with respiratory failure from pneumonia requiring invasive mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | maxiumum of 12 months

SECONDARY OUTCOMES:
Hospital length of stay | maximum of 12 months
ICU length of stay | maximum of 12 months
Days of invasive mechanical ventilation | maximum of 12 months
Total days of antibiotic, antiviral, and antifungal administration (collected both as a total days of therapy and by individual agent) | maximum of 12 months (including planned course of antibiotics to be continued upon discharge)
  The investigators will collect this information by reviewing the electronic medical record which delineates dates and times of each of the medications administered to a participant by nursing staff. The specific dates as well as total consecutive calendar days of each antibiotic administered will be charted in a database for further analysis. Antibiotics will be ranked for spectrum of activity based on microbial coverage as per the Barnes-Jewish Hospital antibiogram most recently published in 2014. De-escalation will be defined as a decrease in number and/or spectrum of antimicrobials administered. Antibiotics, antiviral, antifungals including those which fall into the following classes will be recorded: Penicillins, Floroquinalones, Macrolides, Vancomycin, Linezolid, Cephalosporins, Carbapenems, Monobactams, Aztreonam, Aminoglycocides, Tetracyclines, Metronidazole, non-specific antifungals, Azoles & derivatives, antivirals.
Total days of septic shock as defined by the requirement of vasopressor therapy for maintaining a MAP > 60 | maximum of 12 months
  The electronic medical record will be utilized to determine the number of days for which a participant required vasopressor therapy for blood pressure support. Norepinephrine, Vasopressin, and Phenylephrine are considered vasopressors for this study.
Occurrence of ventilator-associated events | maximum of 12 months
  tracheostomy placement, VAP, pneumothorax while on ventilator
Disposition | maximum of 12 months
  Discharge documentation and social work notes will be reviewed to determine if the patient was discharged to home, an extended care facility/skilled nursing facility, hospice (at home or facility), long term acute care hospital, psychiatric ward, other hospital, or inpatient rehabilitation center. If the patient died in the hospital prior any discharge, this will be documented as the disposition.
90 day readmission rate | 90 days from time of discharge from index hospitalization
  readmission all causes at 90 days post-discharge from index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Marin Kollef, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vidaur L, Planas K, Sierra R, Dimopoulos G, Ramirez A, Lisboa T, Rello J. Ventilator-associated pneumonia: impact of organisms on clinical resolution and medical resources utilization. Chest. 2008 Mar;133(3):625-32. doi: 10.1378/chest.07-2020. Epub 2008 Jan 15. PMID 18198250
- [Background] Kollef MH, Chastre J, Clavel M, Restrepo MI, Michiels B, Kaniga K, Cirillo I, Kimko H, Redman R. A randomized trial of 7-day doripenem versus 10-day imipenem-cilastatin for ventilator-associated pneumonia. Crit Care. 2012 Nov 13;16(6):R218. doi: 10.1186/cc11862. PMID 23148736
- [Background] Chastre J, Fagon JY. Ventilator-associated pneumonia. Am J Respir Crit Care Med. 2002 Apr 1;165(7):867-903. doi: 10.1164/ajrccm.165.7.2105078. PMID 11934711
- [Background] Charlson ME, Sax FL, MacKenzie CR, Fields SD, Braham RL, Douglas RG Jr. Assessing illness severity: does clinical judgment work? J Chronic Dis. 1986;39(6):439-52. doi: 10.1016/0021-9681(86)90111-6. PMID 3086355
- [Background] Dharmarajan K, Hsieh AF, Lin Z, Bueno H, Ross JS, Horwitz LI, Barreto-Filho JA, Kim N, Bernheim SM, Suter LG, Drye EE, Krumholz HM. Diagnoses and timing of 30-day readmissions after hospitalization for heart failure, acute myocardial infarction, or pneumonia. JAMA. 2013 Jan 23;309(4):355-63. doi: 10.1001/jama.2012.216476. PMID 23340637
- [Background] Tang VL, Halm EA, Fine MJ, Johnson CS, Anzueto A, Mortensen EM. Predictors of rehospitalization after admission for pneumonia in the veterans affairs healthcare system. J Hosp Med. 2014 Jun;9(6):379-83. doi: 10.1002/jhm.2184. Epub 2014 Mar 19. PMID 24648401
- [Background] Cabre M, Serra-Prat M, Force L, Almirall J, Palomera E, Clave P. Oropharyngeal dysphagia is a risk factor for readmission for pneumonia in the very elderly persons: observational prospective study. J Gerontol A Biol Sci Med Sci. 2014 Mar;69(3):330-7. doi: 10.1093/gerona/glt099. Epub 2013 Jul 5. PMID 23833199
- [Background] Iregui M, Ward S, Sherman G, Fraser VJ, Kollef MH. Clinical importance of delays in the initiation of appropriate antibiotic treatment for ventilator-associated pneumonia. Chest. 2002 Jul;122(1):262-8. doi: 10.1378/chest.122.1.262. PMID 12114368
- [Background] Micek ST, Lang A, Fuller BM, Hampton NB, Kollef MH. Clinical implications for patients treated inappropriately for community-acquired pneumonia in the emergency department. BMC Infect Dis. 2014 Feb 5;14:61. doi: 10.1186/1471-2334-14-61. PMID 24499035
- [Background] Kollef MH, Shorr A, Tabak YP, Gupta V, Liu LZ, Johannes RS. Epidemiology and outcomes of health-care-associated pneumonia: results from a large US database of culture-positive pneumonia. Chest. 2005 Dec;128(6):3854-62. doi: 10.1378/chest.128.6.3854. PMID 16354854
- [Background] Micek ST, Kollef KE, Reichley RM, Roubinian N, Kollef MH. Health care-associated pneumonia and community-acquired pneumonia: a single-center experience. Antimicrob Agents Chemother. 2007 Oct;51(10):3568-73. doi: 10.1128/AAC.00851-07. Epub 2007 Aug 6. PMID 17682100
- [Background] Shorr AF, Zilberberg MD, Reichley R, Kan J, Hoban A, Hoffman J, Micek ST, Kollef MH. Readmission following hospitalization for pneumonia: the impact of pneumonia type and its implication for hospitals. Clin Infect Dis. 2013 Aug;57(3):362-7. doi: 10.1093/cid/cit254. Epub 2013 May 15. PMID 23677872
- [Background] Magill SS, Klompas M, Balk R, Burns SM, Deutschman CS, Diekema D, Fridkin S, Greene L, Guh A, Gutterman D, Hammer B, Henderson D, Hess D, Hill NS, Horan T, Kollef M, Levy M, Septimus E, VanAntwerpen C, Wright D, Lipsett P. Developing a new, national approach to surveillance for ventilator-associated events*. Crit Care Med. 2013 Nov;41(11):2467-75. doi: 10.1097/CCM.0b013e3182a262db. PMID 24162674
- [Derived] Trupka T, Fisher K, Micek ST, Juang P, Kollef MH. Enhanced antimicrobial de-escalation for pneumonia in mechanically ventilated patients: a cross-over study. Crit Care. 2017 Jul 15;21(1):180. doi: 10.1186/s13054-017-1772-4. PMID 28709439